CLINICAL TRIAL: NCT05475860
Title: Predictors of Atrial High Rate Episodes in Patients Implanting Cardiac Implantable Electronic Device Based on Biomarkers
Brief Title: Biomarkers Predicting Atrial High Rate Episodes in Cardiac Implantable Electronic Device Recipients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Jinhee Ahn, MD, Clinical associate professor, Pusan National University Hospital
Other Study IDs: H-1803
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Atrial High Rate Episode; Cardiac Implantable Electronic Device
MeSH Terms: interventions — Defibrillators, Implantable; Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — biomarkers including soluble ST-2 and FGF-23, single nucleotide polymorphism
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients receiving cardiac implantable electronic device: Patients receiving cardiac implantable electronic device for any clinical indication
  Interventions: Device: implantable cardiac electronic device recipients

INTERVENTIONS:
Device: implantable cardiac electronic device recipients — implantable cardiac electronic device recipients for any clinical indication
  Other Names: pacemaker; implantable cardioverter-defibrillator; cardiac resynchronization therapy

SUMMARY:
This study is sought to investigate any predictors including biomarkers for atrial high rate episodes (AHRE) occurrence in patients without prior history of atrial tachyarrhythmias receiving cardiac implantable electronic device (CIED).

DETAILED DESCRIPTION:
Atrial high rate episodes (AHRE) are noticed up to 70% in patients receiving cardiac implantable electronic device (CIED) even in the absence of prior history of atrial tachyarrhythmias. AHRE is clinically important because it is considered to be associated with clinical atrial fibrillation, stroke, mortality, and heart failure hospitalization. Therefore, predictors of AHRE might be useful for early detection of AHRE susceptable CIED recipients. Biomarkers as well as clinical characteristics will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving cardiac implantable electronic device

Exclusion Criteria:

* patients who disagree for blood sampling to analyze not commonly used clinical biomarkers
* patients not followed-up at least 12 months after implanting device

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving cardiac implantable electronic device for any clinical indication (pacemaker, implantable cardioverter-defibrillator, cardiac resynchronization therapy)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-24 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of atrial high rate episode | 12 months

SECONDARY OUTCOMES:
Factors predicting the occurrence of atrial high rate episode | 12 months
  factors including biomarkers such as FGF-23 and soluble ST-2, and single nucleotide polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Jinhee Ahn, MD, Principal Investigator — Clinical associate professor
Locations (1):
- Jinhee Ahn, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No